CLINICAL TRIAL: NCT03519659
Title: Validating Low FDG Dose PET/CT Compared to Current Standard of Care Dose PET/CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Ohio Third Frontier (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RP0308/2014H0437; R01CA195513 (NIH)
Record Dates: First submitted 2018-02-22; First posted 2018-05-09 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: PET/CT Imaging
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Sub-Study A (Experimental): Patients receive PET/CT scan on Gemini Astonish PET/CT
  Interventions: Diagnostic Test: PET/CT scan with 13 mCi radiation dose; Diagnostic Test: PET/CT scan with 5 mCi radiation dose
- Sub-Study B (Experimental): Patients receive PET/CT scan on Biograph mCT
  Interventions: Diagnostic Test: PET/CT scan with 13 mCi radiation dose; Diagnostic Test: PET/CT scan with 5 mCi radiation dose
- Sub-Study C (Experimental): Patients receive PET/CT scan on Discovery PET/CT
  Interventions: Diagnostic Test: PET/CT scan with 13 mCi radiation dose; Diagnostic Test: PET/CT scan with 5 mCi radiation dose
- Sub-Study D (Experimental): Patients receive PET/CT scan on Vereos 128 digital PET/CT
  Interventions: Diagnostic Test: PET/CT scan with 13 mCi radiation dose; Diagnostic Test: PET/CT scan with 5 mCi radiation dose
- Sub-Study E (Experimental): Patients receive lower radiation dose on Vereos 128 digital PET/CT
  Interventions: Diagnostic Test: PET/CT scan with 2.5 mCi radiation dose; Diagnostic Test: PET/CT Scan with 6.5 mCi radiation dose
- Sub-Study F (Experimental): Patients receive PET/SCAN using system that did not show equivalence in Sub-Study A-C
  Interventions: Diagnostic Test: PET/CT scan with 13 mCi radiation dose; Diagnostic Test: PET/CT Scan with not yet determined radiation dose

INTERVENTIONS:
Diagnostic Test: PET/CT scan with 13 mCi radiation dose — 13 mCi 18F-FDG dose
  Arms: Sub-Study A; Sub-Study B; Sub-Study C; Sub-Study D; Sub-Study F
Diagnostic Test: PET/CT scan with 5 mCi radiation dose — 5 mCi 18F-FDG dose
  Arms: Sub-Study A; Sub-Study B; Sub-Study C; Sub-Study D
Diagnostic Test: PET/CT scan with 2.5 mCi radiation dose — 2.5 mCi 18F-FDG dose
  Arms: Sub-Study E
Diagnostic Test: PET/CT Scan with 6.5 mCi radiation dose — 6.5 mCi 18F-FDG dose
  Arms: Sub-Study E
Diagnostic Test: PET/CT Scan with not yet determined radiation dose — We plan for the possibility that one of the three-Sub-Studies (A-B) would not demonstrate equivalency, and we would then perform a modified protocol in which the SOC dosing is compared to a lower and higher dose than originally tested.
  Arms: Sub-Study F

SUMMARY:
The purpose of this study is to assess new low radiation dose techniques for clinical PET/CT scans through intra-individual comparison between a clinical, standard dose scan and a low-dose scan, completed within one week of each other.

DETAILED DESCRIPTION:
Positron Emission Tomography/Computed Tomography (PET/CT) imaging using 18F-FDG is an important, commonly used cancer, neuroscience and cardio-vascular imaging methodology to detect disease and to monitor therapeutic interventions. While considerable technological progress of PET/CT systems has occurred over the last decade, we have not re-evaluated the ability to potentially reduce the radiation burden of the used PET imaging pharmaceutical (FDG).

This early phase trial intends to accomplish the following:

* to validate that the radiation dose burden from the PET imaging pharmaceutical (FDG) can be reduced by more than 50% from the current standard of clinical care (SOC) level without affecting the diagnostic ability;
* to confirm that a low dose approach will be feasible for response assessment;
* to validate that the difference in FDG uptake between imaging 60 min +/- 10 min post injection and 75 min +/- 10 min post injection is independent/equivalent of the injected FDG dose
* to validate a simulation methodology to streamline future dose finding studies for PET imaging pharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients greater than or equal to 18 years of age
* Patients scheduled for a standard of care PET/CT scan
* For female patients of child-bearing potential, the OSUWMC requirements for receiving the standard of care PET imaging agent and CT examination needs to be met

Exclusion Criteria:

* Participants who are pregnant or lactating
* Prisoners
* Participants incapable of giving informed consent
* Patients unable to lie flat on the scanner for extended periods of time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Image quality | through study completion, on average 2-5 years
  assessed by blinded readers

SECONDARY OUTCOMES:
Artifacts | through study completion, on average 2-5 years
  assessed by blinded readers
Lesion detectability | through study completion, on average 2-5 years
  assessed by blinded readers
Image noise | through study completion, on average 2-5 years
  assessed by blinded readers

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT03519659/Prot_000.pdf